CLINICAL TRIAL: NCT04965935
Title: Efficacy, Mechanisms and Safety of SGLT2 Inhibitors in Kidney Transplant Recipients: The INFINITI Study
Brief Title: Efficacy, Mechanisms and Safety of SGLT2 Inhibitors in Kidney Transplant Recipients
Acronym: INFINITI2019
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sunita Singh, MD, MSc, FRCPC, Clinician Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-5342
Record Dates: First submitted 2021-05-21; First posted 2021-07-16 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant Recipients; Post-transplant Diabetes Mellitus; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Study participants will be allocated to receive either 10 mg daily of dapagliflozin or a matching placebo for 12 weeks in a 1:1 ratio while continuing on existing medical therapy for glycemic control as recommended by Diabetes Canada.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each bottle of drug will be identified with a unique Composite ID in order to maintain the blind. By way of an Unblinding List, Pharmacy will provide treatment allocations of each Composite ID. The Unblinding List will be maintained within a secure location in the Pharmacy. Blinded personnel will not have access to this list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin Tablets (Experimental): Patients will be randomized to therapy with dapagliflozin 10mg PO daily for 12 weeks.
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet
- Placebo Matching Dapagliflozin Tablets (Placebo Comparator): Patients will be randomized to therapy with placebo matching dapagliflozin tablets PO daily for 12 weeks.
  Interventions: Drug: Placebo Matching Dapagliflozin Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 MG Oral Tablet — Dapagliflozin will be administered in a dose of 10 mg/day for 12 weeks.
  Arms: Dapagliflozin Tablets
Drug: Placebo Matching Dapagliflozin Oral Tablet — Placebo will be administered for 12 weeks.
  Arms: Placebo Matching Dapagliflozin Tablets

SUMMARY:
This study will be a randomized, double-blind, placebo-controlled clinical trial comparing the SGLT2 inhibitor dapagliflozin to placebo in 52 kidney transplant recipients (KTR) with or without pre-existing type 2 diabetes (T2D) or post-transplant diabetes mellitus (PTDM). The primary outcome of the trial is to determine if dapagliflozin is superior to placebo in reduction of blood pressure in KTR.

DETAILED DESCRIPTION:
Kidney transplantation is the renal replacement therapy of choice for patients with end stage renal disease (ESRD). It has been well established that kidney transplantation improves patient survival and quality of life, and results in significant savings to the health care system.

Despite the survival benefit conferred by transplantation, KTR still face a number of challenges, especially in patients with diabetes. First, KTR still have a higher risk of mortality than their age-matched counterparts without kidney disease. This mortality risk is even greater amongst KTR with diabetes. Furthermore, mortality from cardiovascular disease (CVD) continues to be an important problem after transplantation. Another major challenge faced by KTR is the continuing risk of developing graft failure over time. Unfortunately, in the subgroup of KTR with diabetes, the incidence of graft failure is 50% higher than the general kidney transplant recipient population, and recurrent diabetic kidney disease (DKD) occurs in almost half of allografts after transplantation. Current strategies in the management of graft dysfunction and chronic kidney disease (CKD) are focused on optimizing immunosuppression and control of hypertension and dyslipidemia. Accordingly, there is an important unmet need for cardio- and renoprotective strategies to address premature death and graft loss in the KTR population.

Sodium-glucose cotransporter 2 inhibitors (SGLT2i) are glucose lowering agents that are effective in the treatment of T2D, resulting not only in improved glycemic control, but also weight loss, blood pressure and albuminuria reduction. Several clinical trials have shown significant benefits of SGLT2i on cardiovascular and renal outcomes. Given the glucose-dependent and independent effects of SGLT2i, as well as the accumulating evidence demonstrating cardiorenal protection in non-KTR, the use of these agents in KTR is attractive - especially since traditional renin-angiotensin-aldosterone system inhibitors are not effective. Moreover, the use of SGLT2i as a cardiorenal protective therapy may be of particular value in KTR given the high burden of comorbidities such as diabetes, CVD and hypertension, as well as the ongoing challenges of premature death and graft loss in this population.

This study will be a randomized, double-blind, placebo-controlled clinical trial comparing the SGLT2 inhibitor dapagliflozin to placebo in 52 KTR with or without pre-existing T2D or PTDM. The primary outcome of the trial is to determine if dapagliflozin is superior to placebo in reduction of blood pressure in KTR. The secondary outcomes of this study include metabolic, vascular, renal and transplant-specific measures. These outcomes have been included to elucidate the potential mechanisms responsible for blood pressure lowering, and putative cardio- and renoprotective effects in KTR. Safety outcomes will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females >18 years old ≥ 6months after kidney transplantation;
2. In patients with T2D or PTDM, HbA1c <12.0%;
3. eGFR ≥30 ml/min/1.73m^2 (as per the CKD-EPI equation);
4. BMI ≤45kg/m^2;
5. Blood pressure ≤160/90 and ≥90/60 at screening.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes;
2. Presence of severe peripheral vascular disease (i.e. prior amputation, gangrene, non-healing ulcer or ischemic rest pain);
3. Presence of acute coronary syndrome, stroke or transient ischemic attack in the 3 months prior to screening;
4. Prior episode of graft pyelonephritis in the 1 month prior to screening;
5. Episode of acute graft rejection in the 3 months prior to screening;
6. Initiation of a new immunosuppressive agent or discontinuation of an immunosuppressive agent in the 1 month prior to screening;
7. Untreated urinary or genital tract infection;
8. Severe hypoglycemia within 3 months of screening, or hypoglycemia unawareness;
9. Pre-menopausal women who are nursing, pregnant, or of child-bearing potential and not practicing an acceptable method of birth control;
10. Participation in another trial with an investigational drug within 30 days of informed consent;
11. Alcohol or drug abuse within 3 months prior to informed consent that would interfere with trial participation;
12. Any ongoing clinical condition that would jeopardize subject safety or study compliance based on investigator judgement.
13. Patients currently using antipsychotic medications.
14. Use of SGLT2 inhibitors within 1 month of starting the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Change from baseline systolic blood pressure (SBP) at 12 weeks of treatment
  SBP

SECONDARY OUTCOMES:
Fasting plasma glucose | Change from baseline fasting plasma glucose at 12 weeks of treatment
  Fasting plasma glucose
HbA1c | Change from baseline HbA1c at 12 weeks of treatment
  HbA1c
Continuous home glucose monitoring | Continuous glucose will be monitored for 14 days at 2 time intervals: 7 days prior to 7 days after drug administration (week -1 to1) and 7 days prior to 7 days after during drug discontinuation (week 11 to 13)
  Continuous home glucose monitoring
Arterial stiffness | Change from baseline arterial stiffness at 12 weeks of treatment
  Measured using a Sphygmocor device
Systemic vascular resistance | Change from baseline systemic vascular resistance at 12 weeks of treatment
  Measured using non-invasive cardiac output monitor (NICOM)
Glomerular Filtration Rate | Change from baseline GFR (based on plasma iohexol clearance) at 12 weeks of treatment
  GFR
Estimated Glomerular Filtration Rate | Change from baseline eGFR (based on CKD-EPI equation) at 12 weeks of treatment
  eGFR
Proximal tubular natriuresis | Change from baseline proximal tubular natriuresis at 12 weeks of treatment
  Measured by fractional excretion of sodium and 24-hour urine collection
Albuminuria | Change from baseline albuminuria at 12 weeks of treatment
  Albuminuria
Urinary and plasma concentration of oxidative stress markers | Change from baseline oxidative stress markers at 12 weeks of treatment
  Measured using ELISA
Tubulointerstitial hypoxia | Change from baseline tubulointerstitial hypoxia at 12 weeks of treatment
  Measured using a renal ultrasound (photoacoustic ultrasonography)
Calcineurin inhibitor (CNI) Levels | Change from baseline CNI at 12 weeks of treatment
  CNI
Adverse Events (AEs) | Adverse events will be recorded from baseline throughout the study duration up to 13 weeks
  AEs

CONTACTS AND LOCATIONS:
Overall Officials: Sunita KS Singh, MD MSc FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Renal Physiology Laboratory, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sridhar VS, Kugathasan L, Lytvyn Y, Liu H, Deng Y, Lovblom LE, Nardone M, Yuen DA, Chen Y, Hua J, Aronson Y, Mohsen M, Kim SJ, Udell JA, Perkins BA, Stevens J, Touw DJ, Heerspink HJL, Cherney DZI, Singh SKS. Efficacy, Mechanisms, and Safety of Sodium-Glucose Cotransporter-2 Inhibitors in Kidney Transplant Recipients: A Randomized, Double-Blind, Placebo-Controlled Trial. Clin J Am Soc Nephrol. 2025 Dec 12. doi: 10.2215/CJN.0000000951. Online ahead of print. No abstract available. PMID 41385300

DOCUMENTS (2):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT04965935/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT04965935/SAP_002.pdf